CLINICAL TRIAL: NCT05988814
Title: Phase II Trial Evaluating the Efficacy and the Safety of FOLFIRINOX3 Treatment in Patients With Unresectable Locally Advanced or Metastatic Pancreatic Cancer in First Line of Chemotherapy (FOLFIRINOX3 Pancréas)
Brief Title: Trial Evaluating the Efficacy and the Safety of FOLFIRINOX3 Treatment in Patients With Unresectable Locally Advanced or Metastatic Pancreatic Cancer in First Line of Chemotherapy
Acronym: FOLFIRINOX3 P
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-505889-29-00
Record Dates: First submitted 2023-07-20; First posted 2023-08-14 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: FOLFIRINOX treatment; pancreatic cancer; first line chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOLFIRINOX treatment (Experimental): Treatment with FOLFIRINOX3 will be administered with a maximum of 16 courses divided into two 8-course doses.
  Maintenance treatment (folinic acid/calcium levofolinate + 5-FU) will be administered until progression.
  Interventions: Drug: FOLFIRINOX treatment

INTERVENTIONS:
Drug: FOLFIRINOX treatment — Treatment with FOLFIRINOX3 will be administered with a maximum of 16 courses divided into two 8-course doses.
  Maintenance treatment (folinic acid/calcium levofolinate + 5-FU) will be administered until progression

SUMMARY:
Evaluate the efficacy of treatment FOLFORINOX 3 in first-line therapy for patients with locally advanced unresectable or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
Evaluate the efficacy of treatment FOLFORINOX 3 in first-line therapy for patients with locally advanced unresectable or metastatic pancreatic cancer.

Treatment with FOLFIRINOX3 will be administered with a maximum of 16 courses divided into two 8-course doses. Maintenance treatment (folinic acid/calcium levofolinate + 5-FU) will be administered until progression.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age > 18 years at time of study entry
* Performance status of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG)
* Patients with pancreatic adenocarcinoma
* Patients with unresectable locally advanced pancreatic cancer or metastatic pancreatic cancer
* Patients with no history of chemotherapy (prior adjuvant or neoadjuvant chemotherapy accepted if the time between the end of chemotherapy and recurrence is greater than 12 months) and no history of curative radiotherapy for metastatic or locally advanced disease. Palliative radiotherapy is accepted.
* Patient eligible for treatment with FOLFIRINOX (5-FU, Irinotecan, Oxaliplatin and folinic acid) including but not limited to: No active heart disease An ECG with a QT/QTc interval ˂ to 450 ms for men and ˂ to 470 ms for women. No uncontrolled hypertension defined by systolic pressure > 140 mmHg or diastolic pressure > 90 mmHg despite optimal medical management. A negative pregnancy test if applicable
* Tumor evaluation (CT scan) performed within 4 weeks (28 days) prior to inclusion with at least one measurable lesion according to RECIST 1.1 criteria
* Patient fit and able to comply with the protocol for the duration of the study, including treatment, visits, scheduled examinations and follow-up.
* Biological, hepatic, renal and serological data within the following limits (tests performed within 7 days of inclusion except for serologies performed within 28 days)
* Information given and informed consent signed
* Patient affiliated to a social security scheme
* Men and women must have an effective contraceptive method.

Exclusion Criteria:

* Patient with neuroendocrine carcinoma or acinar cell carcinoma
* Other cancer in the 5 years preceding inclusion or concomitant (except cancer in situ of the uterine cervix or cutaneous basal cell carcinoma).
* Presence of brain metastasis(es)
* Estimated prognosis < 3 months
* History of grade 4 toxicity to oxaliplatin, irinotecan or 5FU if history of adjuvant/neoadjuvant chemotherapy
* Sequellar toxicity > grade 1 if previous adjuvant/neoadjuvant chemotherapy
* Hypersensitivity to any component of FOLFIRINOX® treatment.
* Current participation or participation within 30 days prior to inclusion in another therapeutic trial with an investigational compound and/or completion of radiotherapy within 10 days prior to the start of treatment
* Evidence of a homozygous or heterozygous DPYD mutation and/or uracilemia >16ng/mL and/or homozygous UGT1A1 genotype.
* Pregnancy, breastfeeding
* Inability to sign informed consent or to undergo medical monitoring of the trial for geographical, social or psychological reasons including, but not limited to, psychiatric illness compromising comprehension of information or conduct of the study.
* Patient under guardianship, curatorship or safeguard of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2029-07-24 (Estimated); Study Completion 2029-07-24 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 6 months
  Progression-free survival (PFS) on FOLFIRINOX3 at 6 months.

SECONDARY OUTCOMES:
Overall survival (OS) | 24 months
  Overall survival (OS) is defined as the time interval between the date of inclusion and the date of death from any cause.
Acute and late toxicities (adverses events) | Until 30 days after the end of treatment
  Acute toxicity is defined as toxicity occurring within 6 months of the start of chemotherapy.
  A toxicity is late if it occurs more than 6 months after the start of chemotherapy.
Quality of life (QoL) | Until the end of treatment an average of 14 months
  Quality of life (QoL) will be assessed at inclusion, every 4 courses up to 6 months, then every 8 courses using questionnaires validated by the EORTC (European Organisation for Research and Treatment of Cancer): the cancer-specific QLQ-C30
Quality of life (QoL) | Until the end of treatment an average of 14 months
  Quality of life (QoL) will be assessed at inclusion, every 4 courses up to 6 months, then every 8 courses using questionnaires validated by the EORTC (European Organisation for Research and Treatment of Cancer): the QLQPAN26,a module specific to pancreatic cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Georges-François Leclerc, Dijon, France